CLINICAL TRIAL: NCT02808533
Title: Topiramate in Treatment Refractory Psychotic Illness: Effects on Weight Gain and Psychopathology
Brief Title: Topiramate and Schizophrenia: Effects on Weight and Psychopathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Margaret Hahn, Clinician-Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 097/2015
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia, Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate (Experimental): Topiramate will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): Placebo will be dispensed on a biweekly basis, and pill counts conducted at each visit.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate capsules starting with 25 mg b.i.d with an incremental increase of 25 mg b.i.d weekly upto a maximum of 100 mg b.i.d.
  Other Names: Topamax
  Arms: Topiramate
Other: Placebo — Placebo capsules visually identical to those containing topiramate will be administered.
  Arms: Placebo

SUMMARY:
Clozapine is the sole AP agent with superiority in treatment refractory schizophrenia, but it also is associated with the greatest risk of weight gain and other metabolic abnormalities. Topiramate, an anticonvulsant agent, possesses a weight-reducing effect. Furthermore, some studies have suggested that Topiramate may be associated with improvements in psychopathology in treatment refractory schizophrenia. Here the investigators propose to determine the role of topiramate for augmentation purposes (psychopathology) and as an adjunctive pharmacological intervention for weight loss in overweight/obese individuals with Ultra-Treatment Resistant Schizophrenia or Schizoaffective disorder taking clozapine.

DETAILED DESCRIPTION:
Schizophrenia is a chronic illness characterized by social and vocational disruptive functioning. While >70% of individuals with first episode illness respond to antipsychotics (APs), there remains a subgroup left with persisting psychotic symptoms. For these individuals, clozapine (CLZ) is also the sole drug with treatment superiority, but also carries the greatest metabolic liability. Another complicating factor in those treated with CLZ is the observation that while effective in some, 40-70% of individuals fail to show significant improvement with CLZ, often leading to augmentation strategies. While controlled trials are, in general lacking, a number of agents have been suggested as useful. One such group of medications includes the anticonvulsants.

Topiramate represents one of the newer anticonvulsant agents approved for the treatment of epilepsy and prophylaxis of migraines. Importantly, topiramate possesses a weight-reducing effect that has been substantiated by a meta-analysis in non-psychiatric patients. Interestingly, topiramate has been studied as an adjunctive therapy in treatment-resistant schizophrenia with some evidence demonstrating small to moderate benefits with topiramate augmentation on psychopathology. However, these benefits must also be weighed against reports (primarily from epilepsy populations), that topiramate may cause cognitive dysfunction.

This study will examine:

1. Topiramate-related effects on weight
2. Topiramate-related effects on glucose tolerance and insulin sensitivity
3. Topiramate-related effects on psychopathology and cognition
4. Topiramate-related effects on adiposity

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Schizoaffective disorder
* 17-59 years of age
* Clozapine treatment for at least 12 weeks at a dose 350 mg/d or greater and/or plasma clozapine levels of 300 ng/mL or greater
* CGI must be 4 or higher and/or GAF < 50
* BMI greater than or equal to 25

Exclusion Criteria:

* Alcohol use disorder
* Patients with liver, or renal dysfunction
* Females of child bearing age not on a regular contraceptive, females who are nursing
* Clinical or laboratory evidence of uncompensated cardiovascular, endocrine, hematological, or pulmonary disease.
* HbA1c > 9%, or symptomatic hyperglycemia with metabolic decompensation
* Prior lack of efficacy or tolerability of Topiramate
* Addition of new hypoglycemic or lipid lowering medication within 2 months of starting study
* Patients treated with Valproic Acid
* Patients treated with hydrochlorothiazide
* Switch in antipsychotic medications within 3 months of study entry
* Major medical or surgical event within the preceding 3 months
* History of renal stones
* Use of Carbonic Anhydrase Inhibitor
* History of glaucoma
* Acute Suicidal risk

Ages: 17 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 16 weeks
  Measured in pounds

SECONDARY OUTCOMES:
Insulin sensitivity | 16 weeks
  Measured through Oral Glucose Tolerance Test (pmol/L)
Psychopathology - Positive and Negative Syndrome Scale (PANSS) | 16 weeks
  Anchored scale to rate positive and negative psychiatric symptoms
Glucose Tolerance | 16 weeks
  Measured through Oral Glucose Tolerance Test (mmol/L)
Psychopathology - Brief Psychiatric Rating Scale (BPRS) | 16 weeks
  Anchored rating scale for psychiatric symptoms
Psychopathology - Clinical Global Impression (CGI) | 16 weeks
  Anchored scale to rate global impression of patient
Psychopathology - Global Assessment of Functioning (GAF) | 16 weeks
  Anchored scale to rate global functioning of patient

OTHER OUTCOMES:
Visceral adiposity changes | Baseline and 16 weeks
  Measured through MRI
Cognition - Brief Assessment of Cognition in Schizophrenia (BACS) | 16 weeks
  A standardized assessment of cognitive in patients with schizophrenia
Volumetric Brain changes | Baseline and 16 weeks
  Measured through MRI
Hepatic adiposity changes | Baseline and 16 weeks
  Measured through MRI

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hahn, PhD, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research